CLINICAL TRIAL: NCT04603781
Title: Use of CBD Oil for Reducing the Negative Emotional Impact of COVID-19: A Randomized Placebo-Controlled Clinical Trial
Brief Title: CBD Oil for Reducing Emotional Impact of COVID-19
Acronym: CBDOIL
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Suspended (The UT IRB determined that CBD oil is being used as a drug as defined by the FDA. Therefore, an IND must be obtained for the use of CBD oil in this research study in accordance with FDA regulations, 21 CFR 312.)
Sponsor: University of Texas at Austin (Other)
Collaborators: Way West Wellness (Unknown); SunFlora.Inc (Unknown)
Responsible Party: Principal Investigator, Michael J. Telch, Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-07-0138
Record Dates: First submitted 2020-10-03; First posted 2020-10-27 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Anxiety Depression; Alcohol Abuse; Substance Abuse; Anger; Sleep Disturbance; Stress Reaction
Keywords: CBD Oil; CBD Isolate; COVID-19; stress symptoms; RCT
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Parasomnias; Fractures, Stress; COVID-19

STUDY DESIGN:
Intervention Model Description: 4-arm double-blind placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The PI and all members of the study team will be blind to the drug assignment of the patient. Only the CBD suppliers (John Fornecker- Way West and Anthony Ferrari - SunMed CBD) and a UT LSAD staff member (not connected to the study) will have access to participants' treatment assignment. In the very unlikely event that a participant should have an adverse reaction requiring medical attention, the PI will contact the UT staff person who is keeper of the blind and request the treatment assignment of the subject in question without revealing the treatment condition coding scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CBD-Isolate 300 mg. (Active Comparator): Nightly oral administration of 300 mg. of CBD-Isolate for 28 consecutive days
  Interventions: Dietary Supplement: CBD Isolate
- Full-Spectrum CBD Oil 300 mg. (Active Comparator): Nightly oral administration of 300 mg. of Full Spectrum CBD Oil for 28 consecutive days
  Interventions: Dietary Supplement: Full Spectrum CBD Oil
- Broad-Spectrum CBD oil 300 mg. (Active Comparator): Nightly oral administration of 300 mg. of Broad-Spectrum CBD Oil for 28 consecutive days
  Interventions: Dietary Supplement: Broad-Spectrum CBD Oil
- Placebo Oil (Placebo Comparator): Nightly oral administration of 300 mg. of Placebo Oil for 28 consecutive days
  Interventions: Dietary Supplement: Placebo Oil

INTERVENTIONS:
Dietary Supplement: CBD Isolate — 300 mg. daily dose of CBD Isolate Oil
  Other Names: Pure CBD oil
  Arms: CBD-Isolate 300 mg.
Dietary Supplement: Full Spectrum CBD Oil — 300 mg. daily dose of CBD with full spectrum of other cannabinoids found in the hemp plant
  Arms: Full-Spectrum CBD Oil 300 mg.
Dietary Supplement: Broad-Spectrum CBD Oil — 300 mg. daily dose of CBD with a selected spectrum of other cannabinoids found in the hemp plant
  Arms: Broad-Spectrum CBD oil 300 mg.
Dietary Supplement: Placebo Oil — MCT Oil with mint flavoring
  Arms: Placebo Oil

SUMMARY:
Our purpose is to conduct a 4-arm placebo-controlled clinical trial to investigate the relative clinical efficacy of 300 mg. of pure hemp-derived CBD isolate, 300 mg. of full spectrum CBD oil, 300 mg. of broad- spectrum CBD Oil, or Placebo oil among adults presenting with COVID-19 -induced stress reactions including one or more of the following: anxiety, depression, anger, substance use, or sleep disturbance.

DETAILED DESCRIPTION:
Background and Significance of the Proposed Project

The COVID-19 pandemic has hit us like a ton of bricks creating unimaginable levels of unanticipated death, financial hardship, and dramatic changes in nearly every facet of our life including school, work, shopping, social and family life. Sadly, the physical, mental, economic, and health burden of COVID-19 disproportionately affects the poor, the elderly, and people of color.

The stress induced by these changes as well as the lack of control we have over them increases risk for new onset of mental health problems such as anxiety, depression, substance abuse, sleep disturbance, and family violence as well as exacerbation of symptoms among those with pre-existing psychiatric conditions. Although many people will successfully manage the increased stress from COVID-19 on their own or with the support from family and friends, others may need extra help to cope. Consequently, there is an urgent need for developing cost-effective strategies for managing the stress-induced psychological consequences of COVID-19.

There's been considerable excitement in the press over the potential therapeutic use of cannabidiol (CBD) products in the treatment of a variety of physical and mental health problems. Delta-9-tetrahydrocannabinol (delta-9 THC) is still illegal in most states because of its psychoactive abuse potential. In contrast, cannabidiol (CBD) does not convert to THC in the body and has negligible side effects relative to main-stream psychiatric drugs (benzodiazepines and antidepressants) commonly prescribed for the treatment of stress-related disorders such as anxiety, depression, and insomnia. Mounting evidence from studies with rodents suggests that CBD may confer significant promising health-related benefits including anti-inflammatory, pain-relieving, anti-cancer, memory enhancement, and facilitation of fear extinction (see White for a recent review).

The biggest success story for CBD use in humans to date comes from placebo-controlled randomized clinical trials demonstrating a 50% or more reduction in previously intractable seizures in children suffering from Dravet syndrome and Lennox-Gastaut syndrome. Moreover, several controlled clinical trials have shown promising findings in reducing psychotic symptoms among patients with schizophrenia and among young adults displaying THC-induced psychosis.

Preliminary Evidence that CBD may offer promise in the treatment of stress-related disorders has started to emerge. A small pilot trial with 24 patients presenting with social anxiety disorder found that relative to placebo, a single dose of 100 mg of CBD oil led to lower levels of anxiety, cognitive impairment, and discomfort in their actual speech performance as well as their anxiety before the speech. An uncontrolled case series of 11 PTSD patients receiving 8 weeks of CBD, reported a 28% reduction in PTSD symptom scores. In a small 4-week placebo-controlled study of 37 young Japanese adults with social anxiety disorder, Masataka found a significant advantage of CBD over placebo in reducing subjects' scores on two widely used measures of social anxiety symptoms.

Why Compare CBD-Isolate with Broad-Spectrum and Full-Spectrum CBD? CBD isolate is the purest form of CBD. It is made by extracting it from its natural environment - either hemp which is legal and recognized as generally safe in all states because of its low THC content (less than .3%), or the marijuana plant which has high levels of THC (up to 30%) and remains a Schedule 1 controlled substance under the Controlled Substances Act of 1970.

Unlike hemp-derived CBD Isolate, hemp-derived full-spectrum CBD contains all the hundreds of phytochemicals naturally found in the cannabis plant, including CBD, trace cannabinoids including Cannabinol (CBN), Cannabichromene (CBC), Cannabigerol (CBDA) and Cannabidivarin (CBDV), and more than 200 different terpenes, essential oils, and negligible THC content (less than 0.3%).

Research demonstrating the wide-ranging therapeutic effects of CBD oil including anti-emetic, anti-inflammatory, anxiolytic, and anti-psychotic effects were based on studies using pure doses of CBD Isolate. However, more recently it has been shown that the therapeutic effects of purified CBD display a bell-shaped dose-response curve suggesting a limited dose range, with no beneficial effects achieved at either lower or higher doses. This narrow therapeutic window presents a challenge for using CBD isolate clinically.

Based on recent research with rodents and humans, administration of a full spectrum cannabis extract containing mostly CBD but also containing other minor phytocannabinoids and non-cannabinoids exerted a synergistic effect with CBD that was both more effective than CBD Isolate without the unwanted bell-shaped dose-response curve. This finding has been named the entourage effect. However, to date, there are no human trials for any physical or mental health problem comparing the gold standard CBD isolate with a full-spectrum CBD formulation, despite the fact that both forms of CBD are widely available without a prescription in stores all across the United States. The proposed project will provide important data to determine whether a full-spectrum CBD formulation offers any advantages over CBD isolate in reducing COVID-19 stress-induced symptoms.

Specific Aims and Hypotheses:

1. Compare the efficacy of a 4-week daily regimen of hemp-derived CBD isolate (300 mg/day), broad-spectrum CBD oil, full spectrum CBD oil (300 mg/day), or placebo oil in reducing patient-rated symptoms of stress, anxiety, depression, and sleep disturbance. It is predicted that patients receiving and of the three active CBD oil formulations (pure isolate, broad-spectrum, or full spectrum CBD oil) will show significantly greater reduction in emotional distress and sleep disturbance relative to those receiving placebo oil. It is also predicted that broad-spectrum and full-spectrum CBD oil will outperform CBD isolate in reducing COVID-19 stress-induced symptoms of stress, anxiety, depression, anger, and sleep disturbance.
2. Examine predictors of patients' clinical response to the 4 treatments. It is expected that the superiority of broad-spectrum and full-spectrum CBD oil relative to CBD isolate or placebo will be more pronounced for patients showing more severe COVID-19 stress-induced symptoms at baseline.
3. Examine the perceived acceptability and side effects profile of 4 weeks of daily CBD/Placebo oil ingestion. It is expected that each of the three CBD formulations (CBD isolate, Broad-spectrum or Full spectrum CBD oil) will show minimal side effects that will not exceed the level of side effects for those ingesting placebo oil with the possible exception of somnolence.

ELIGIBILITY:
INCLUSION CRITERIA:

* Displays elevated symptom scores on one or more of the following established assessment instruments for depression (PROMIS-Depression), anxiety (PROMIS-Anxiety), Anger (PROMIS-Anger), sleep disturbance (PROMIS-Sleep); or Alcohol/Substance (PROMIS-Alcohol; PROMIS- Substance Use)
* Age between 18 to 70;
* Fluent in English;
* Has home access to the Internet;
* Willingness to provide signed informed consent;
* Willingness to refrain from all non-study CBD products during the 6-week study period;
* Willing to complete a brief pre-study 7-day online symptom monitoring log;
* Currently residing in the United States

EXCLUSION CRITERIA:

* History of a suicide attempt within the past 6 months
* Any medical problem that would preclude participating in the study including liver disease
* Current use of warfarin or other prescribed blood thinners,
* Currently taking seizure medications such as valproate, lamotrigine, or clobazam;
* Currently taking thyroid medications such as levothyroxine;
* Currently taking heart rhythm medications such as amiodarone;
* Currently taking anti-hypertension medications;
* Pregnant or planning to become pregnant within the next 6 weeks.
* History of adverse reaction to CBD oil or other CBD products.
* Allergic to coconut oil.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS Emotional Distress Index | Week 0-Baseline
  This measure is a 43-item patient-rated emotional distress symptom scale consisting of 6 sub-factors (Depression, Anxiety, Anger, Alcohol Use, Substance Use, and Sleep Disturbance). Each symptom is rated over a 7-day period on a 5-point scale.
PROMIS Emotional Distress Index | Week 1-Treatment
  This measure is a 43-item patient-rated emotional distress symptom scale consisting of 6 sub-factors (Depression, Anxiety, Anger, Alcohol Use, Substance Use, and Sleep Disturbance). Each symptom is rated over a 7-day period on a 5-point scale.
PROMIS Emotional Distress Index | Week 2-Treatment
  This measure is a 43-item patient-rated emotional distress symptom scale consisting of 6 sub-factors (Depression, Anxiety, Anger, Alcohol Use, Substance Use, and Sleep Disturbance). Each symptom is rated over a 7-day period on a 5-point scale.
PROMIS Emotional Distress Index | Week 3-Treatment
  This measure is a 43-item patient-rated emotional distress symptom scale consisting of 6 sub-factors (Depression, Anxiety, Anger, Alcohol Use, Substance Use, and Sleep Disturbance). Each symptom is rated over a 7-day period on a 5-point scale.
PROMIS Emotional Distress Index | Week 4-Treatment
  This measure is a 43-item patient-rated emotional distress symptom scale consisting of 6 sub-factors (Depression, Anxiety, Anger, Alcohol Use, Substance Use, and Sleep Disturbance). Each symptom is rated over a 7-day period on a 5-point scale.
PROMIS Emotional Distress Index | Week 5-Follow-up
  This measure is a 43-item patient-rated emotional distress symptom scale consisting of 6 sub-factors (Depression, Anxiety, Anger, Alcohol Use, Substance Use, and Sleep Disturbance). Each symptom is rated over a 7-day period on a 5-point scale.

SECONDARY OUTCOMES:
PROMIS Depression Scale | Week 0-Baseline
  This measure is an 8-item patient-rated depression symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Depression Scale | Week 1-Treatment
  This measure is an 8-item patient-rated depression symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Depression Scale | Week 2-Treatment
  This measure is an 8-item patient-rated depression symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Depression Scale | Week 3-Treatment
  This measure is an 8-item patient-rated depression symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Depression Scale | Week 4-Treatment
  This measure is an 8-item patient-rated depression symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Depression Scale | Week 5-Follow-up
  This measure is an 8-item patient-rated depression symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Anxiety Scale | Week 0- Baseline
  This measure is an 8-item patient-rated anxiety symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Anxiety Scale | Week 1-Treatment
  This measure is an 8-item patient-rated anxiety symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Anxiety Scale | Week 2-Treatment
  This measure is an 8-item patient-rated anxiety symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Anxiety Scale | Week 3-Treatment
  This measure is a 7-item patient-rated anxiety symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Anxiety Scale | Week 4-Treatment
  This measure is a 7-item patient-rated anxiety symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Anxiety Scale | Week 5-Follow-up
  This measure is a 7-item patient-rated anxiety symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Anger Scale | Week 0- Baseline
  This measure is a 5-item patient-rated anger symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Anger Scale | Week 1- Treatment
  This measure is a 5-item patient-rated anger symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Anger Scale | Week 2- Treatment
  This measure is a 5-item patient-rated anger symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Anger Scale | Week 3- Treatment
  This measure is a 5-item patient-rated anger symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Anger Scale | Week 4- Treatment
  This measure is a 5-item patient-rated anger symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Anger Scale | Week 5- Follow-up
  This measure is a 5-item patient-rated anger symptom scale. Each symptom is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Alcohol Negative Consequences Scale | Week 0- Baseline
  This measure is a 7-item patient-rated index of alcohol-related problems. Each item is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Alcohol Negative Consequences Scale | Week 1- Treatment
  This measure is a 7-item patient-rated index of alcohol-related problems. Each item is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Alcohol Negative Consequences Scale | Week 2- Treatment
  This measure is a 7-item patient-rated index of alcohol-related problems. Each item is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Alcohol Negative Consequences Scale | Week 3- Treatment
  This measure is a 7-item patient-rated index of alcohol-related problems. Each item is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Alcohol Negative Consequences Scale | Week 4- Treatment
  This measure is a 7-item patient-rated index of alcohol-related problems. Each item is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Alcohol Negative Consequences Scale | Week 5- Follow-up
  This measure is a 7-item patient-rated index of alcohol-related problems. Each item is rated over a 7-day period on a 5-point scale ranging from 1 (Never) to 5 (Always).
PROMIS Sleep Disturbance Scale | Week 0- Baseline
  This measure is an 8-item patient-rated index of sleep disturbance. Each item is rated over a 7-day period on a 5-point scale ranging from 1 (Not at all) to 5 (Very Much).
PROMIS Sleep Disturbance Scale | Week 1- Treatment
  This measure is an 8-item patient-rated index of sleep disturbance. Each item is rated over a 7-day period on a 5-point scale ranging from 1 (Not at all) to 5 (Very Much).
PROMIS Sleep Disturbance Scale | Week 2- Treatment
  This measure is an 8-item patient-rated index of sleep disturbance. Each item is rated over a 7-day period on a 5-point scale ranging from 1 (Not at all) to 5 (Very Much).
PROMIS Sleep Disturbance Scale | Week 3- Treatment
  This measure is an 8-item patient-rated index of sleep disturbance. Each item is rated over a 7-day period on a 5-point scale ranging from 1 (Not at all) to 5 (Very Much).
PROMIS Sleep Disturbance Scale | Week 4- Treatment
  This measure is an 8-item patient-rated index of sleep disturbance. Each item is rated over a 7-day period on a 5-point scale ranging from 1 (Not at all) to 5 (Very Much).
PROMIS Sleep Disturbance Scale | Week 5- Follow-up
  This measure is an 8-item patient-rated index of sleep disturbance. Each item is rated over a 7-day period on a 5-point scale ranging from 1 (Not at all) to 5 (Very Much).
COVID-19 Coping Self-Efficacy | Week 0- Baseline
  This measure is a 15-item author-constructed patient-rated index of COVID-19 Coping Self-Efficacy
COVID-19 Coping Self-Efficacy | Week 1- Treatment
  This measure is a 15-item author-constructed patient-rated index of COVID-19 Coping Self-Efficacy
COVID-19 Coping Self-Efficacy | Week 2- Treatment
  This measure is a 15-item author-constructed patient-rated index of COVID-19 Coping Self-Efficacy
COVID-19 Coping Self-Efficacy | Week 3- Treatment
  This measure is a 15-item author-constructed patient-rated index of COVID-19 Coping Self-Efficacy
COVID-19 Coping Self-Efficacy | Week 4- Treatment
  This measure is a 15-item author-constructed patient-rated index of COVID-19 Coping Self-Efficacy
COVID-19 Coping Self-Efficacy | Week 5- Follow-up
  This measure is a 15-item author-constructed patient-rated index of COVID-19 Coping Self-Efficacy
Sheehan Disability Scale | Week 0- Baseline
  This measure is a 3-item patient-rated index of level of functional impairment.
Sheehan Disability Scale | Week 5- Follow-up
  This measure is a 3-item patient-rated index of level of functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Telch, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Laboratory for the Study of Anxiety Disorders, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cowger TL, Davis BA, Etkins OS, Makofane K, Lawrence JA, Bassett MT, Krieger N. Comparison of Weighted and Unweighted Population Data to Assess Inequities in Coronavirus Disease 2019 Deaths by Race/Ethnicity Reported by the US Centers for Disease Control and Prevention. JAMA Netw Open. 2020 Jul 1;3(7):e2016933. doi: 10.1001/jamanetworkopen.2020.16933. PMID 32721026
- [Background] Mazza C, Ricci E, Biondi S, Colasanti M, Ferracuti S, Napoli C, Roma P. A Nationwide Survey of Psychological Distress among Italian People during the COVID-19 Pandemic: Immediate Psychological Responses and Associated Factors. Int J Environ Res Public Health. 2020 May 2;17(9):3165. doi: 10.3390/ijerph17093165. PMID 32370116
- [Background] White CM. A Review of Human Studies Assessing Cannabidiol's (CBD) Therapeutic Actions and Potential. J Clin Pharmacol. 2019 Jul;59(7):923-934. doi: 10.1002/jcph.1387. Epub 2019 Feb 7. PMID 30730563
- [Background] Devinsky O, Cross JH, Laux L, Marsh E, Miller I, Nabbout R, Scheffer IE, Thiele EA, Wright S; Cannabidiol in Dravet Syndrome Study Group. Trial of Cannabidiol for Drug-Resistant Seizures in the Dravet Syndrome. N Engl J Med. 2017 May 25;376(21):2011-2020. doi: 10.1056/NEJMoa1611618. PMID 28538134
- [Background] Devinsky O, Patel AD, Cross JH, Villanueva V, Wirrell EC, Privitera M, Greenwood SM, Roberts C, Checketts D, VanLandingham KE, Zuberi SM; GWPCARE3 Study Group. Effect of Cannabidiol on Drop Seizures in the Lennox-Gastaut Syndrome. N Engl J Med. 2018 May 17;378(20):1888-1897. doi: 10.1056/NEJMoa1714631. PMID 29768152
- [Background] McGuire P, Robson P, Cubala WJ, Vasile D, Morrison PD, Barron R, Taylor A, Wright S. Cannabidiol (CBD) as an Adjunctive Therapy in Schizophrenia: A Multicenter Randomized Controlled Trial. Am J Psychiatry. 2018 Mar 1;175(3):225-231. doi: 10.1176/appi.ajp.2017.17030325. Epub 2017 Dec 15. PMID 29241357
- [Background] Zuardi AW, Hallak JE, Dursun SM, Morais SL, Sanches RF, Musty RE, Crippa JA. Cannabidiol monotherapy for treatment-resistant schizophrenia. J Psychopharmacol. 2006 Sep;20(5):683-6. doi: 10.1177/0269881106060967. Epub 2006 Jan 9. PMID 16401651
- [Background] Morgan CJ, Curran HV. Effects of cannabidiol on schizophrenia-like symptoms in people who use cannabis. Br J Psychiatry. 2008 Apr;192(4):306-7. doi: 10.1192/bjp.bp.107.046649. PMID 18378995
- [Background] Bergamaschi MM, Queiroz RH, Chagas MH, de Oliveira DC, De Martinis BS, Kapczinski F, Quevedo J, Roesler R, Schroder N, Nardi AE, Martin-Santos R, Hallak JE, Zuardi AW, Crippa JA. Cannabidiol reduces the anxiety induced by simulated public speaking in treatment-naive social phobia patients. Neuropsychopharmacology. 2011 May;36(6):1219-26. doi: 10.1038/npp.2011.6. Epub 2011 Feb 9. PMID 21307846
- [Background] Elms L, Shannon S, Hughes S, Lewis N. Cannabidiol in the Treatment of Post-Traumatic Stress Disorder: A Case Series. J Altern Complement Med. 2019 Apr;25(4):392-397. doi: 10.1089/acm.2018.0437. Epub 2018 Dec 13. PMID 30543451
- [Background] Masataka N. Anxiolytic Effects of Repeated Cannabidiol Treatment in Teenagers With Social Anxiety Disorders. Front Psychol. 2019 Nov 8;10:2466. doi: 10.3389/fpsyg.2019.02466. eCollection 2019. PMID 31787910
- [Background] Linares IM, Zuardi AW, Pereira LC, Queiroz RH, Mechoulam R, Guimaraes FS, Crippa JA. Cannabidiol presents an inverted U-shaped dose-response curve in a simulated public speaking test. Braz J Psychiatry. 2019 Jan-Feb;41(1):9-14. doi: 10.1590/1516-4446-2017-0015. Epub 2018 Oct 11. PMID 30328956
- [Background] Gallily R, Yekhtin Z, Hanuš LO. Overcoming the Bell-Shaped Dose-Response of Cannabidiol by Using <i>Cannabis</i> Extract Enriched in Cannabidiol. Pharmacol Amp Pharm. 2015;06(02):75-85. doi:10.4236/pp.2015.62010
- [Background] Russo EB. Taming THC: potential cannabis synergy and phytocannabinoid-terpenoid entourage effects. Br J Pharmacol. 2011 Aug;163(7):1344-64. doi: 10.1111/j.1476-5381.2011.01238.x. PMID 21749363